CLINICAL TRIAL: NCT07216612
Title: Recovery Works - Facilitating Sustainable Recovery Through Workforce
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Collaborators: West Virginia First Foundation, Inc. (Unknown)
Responsible Party: Principal Investigator, Brian Hendricks, Principal Investigator, West Virginia School of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R043025BH
Record Dates: First submitted 2025-09-17; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Workforce; Substance Use Disorder; Rural communities
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Day Report employment model (Active Comparator): Participants assigned to the Standard Employment Model will receive cognitive behavioral therapy (CBT) supports offered through the Day Report Program. CBT incorporates small rewards such as gift cards, small giveaways, or hosted events, determined by Day Report case coordinators as part of standard programming. Participants may also be offered the opportunity to enroll in Jobs and Hope West Virginia, a recovery-oriented employment agency that provides support for employees in recovery and employers hiring a recovery workforce. Enrollment in Jobs and Hope WV is encouraged but voluntary. All participants will also have access to free public transportation through the Mountain Transit Authority to commute to and from work.
  Interventions: Other: Standard Employment Model
- CRAFT Workforce Model (Experimental): Participants assigned to the Community Restitution Apprenticeship-Focused Training (CRAFT) workforce model will complete community service assignments focused on job-specific training, participate in apprenticeship-based work experiences with local employers, and receive mentoring from study staff and workplace supervisors. Participants will also maintain routine follow-up with their Day Report Program case managers. The CRAFT model is designed to integrate employment-based skill-building with structured recovery support to improve recovery capital, social capital, and reduce Day Report Program violations.
  Interventions: Other: Community Restitution Apprenticeship-Focused Training (CRAFT)

INTERVENTIONS:
Other: Community Restitution Apprenticeship-Focused Training (CRAFT) — Twenty-five participants will be randomly assigned to the intervention arm. Participants will receive the standard services of the Day Report Program plus enrollment in the CRAFT model. CRAFT involves completion of community service activities designed to develop career-related skills and placement in an apprenticeship with a local employer. Participants may also be offered the opportunity to enroll in Jobs and Hope West Virginia, a recovery-oriented employment program that supports individuals in recovery and employers hiring a recovery workforce. Enrollment in Jobs and Hope WV is encouraged but voluntary.
  Arms: CRAFT Workforce Model
Other: Standard Employment Model — Twenty-five participants will be randomly assigned to the comparator arm. Participants will receive the standard services of the Day Report Program, which include cognitive behavioral therapy (CBT) supports with small incentives such as gift cards, small giveaways, or hosted events determined by Day Report Program case coordinators. Participants may also be offered the opportunity to enroll in Jobs and Hope West Virginia, a recovery-oriented employment program that provides workforce support for individuals in recovery and employers. Enrollment in Jobs and Hope WV is encouraged but voluntary. All participants will also have access to free public transportation through the Mountain Transit Authority to commute to and from work.
  Arms: Standard Day Report employment model

SUMMARY:
The goal of this clinical trial is to determine whether an apprenticeship-based workforce model, the Community Restitution Apprenticeship-Focused Training (CRAFT), improves recovery outcomes for persons with substance use disorder. The main research questions are:

* Does the CRAFT workforce model improve recovery and social capital for justice-involved adults with substance use disorder?
* Does the CRAFT workforce model reduce Day Report Program violations for justice-involved adults with substance use disorder?

Secondary research questions include:

* Are there differences in program effects between men and women?
* Are there differences in program effects across age groups? Researchers will compare the CRAFT apprenticeship-based workforce model to the standard employment model for Day Report Program participants to determine whether the apprenticeship-based model improves outcomes.

Participants assigned to the CRAFT apprenticeship-based workforce model will:

* Complete community service focused on job-specific training
* Meet with study staff monthly to complete questionnaires
* Work with study staff to engage in workplace mentoring
* Maintain consistent follow-up with their Day Report Program case managers

DETAILED DESCRIPTION:
Human Subjects Involvement, Characteristics, and Design This study is a randomized, parallel-arm clinical trial with no blinding, designed to assess the effects of the Community Restitution Apprenticeship-Focused Training (CRAFT) workforce model on recovery and community reintegration outcomes.

Primary outcomes are:

1. Change in social recovery capital score as measured by the REC-CAP Social Recovery Capital Scale
2. Change in personal recovery capital score as measured by the REC-CAP Recovery Capital Index
3. Number of Greenbrier County Day Report Program violations as recorded by case coordinators All outcomes will be assessed over 6 months. Secondary outcomes include analyses of sex-based and age-based differences in recovery capital scores and Greenbrier County Day Report Program (hereinafter referred to as "Day Report Program"), violations over the same 6-month period.

Fifty participants will be recruited from the Day Report Program, a community corrections program located in Greenbrier County, West Virginia. Participants must be ≥18 years of age, actively enrolled in the Day Report Program, and charged with a nonviolent felony or misdemeanor offense with a substance use problem.

Exclusion criteria include:

* Under 18 years of age
* Not enrolled in the Day Report Program
* A prior felony conviction involving the use of force with intent to cause serious bodily harm or death
* A sexual offense
* An offense involving a child victim
* An offense involving the illegal use of a firearm or other dangerous weapon
* Death or serious bodily injury to another person during the commission of the crime
* The use of force against another person during the commission of the crime Recruitment will occur through flyers posted within the Greenbrier County Day Report Center (herafter referred to as "Day Report Center"), referrals from Day Report Program case managers, and a WVSOM Institutional Review Board (IRB)-approved recruitment video presented to potential participants at the Day Report Center. Following referral, study staff will meet with interested clients (and, if applicable, their case manager) to explain the study and begin the informed consent process.

The informed consent process will be conducted using a standardized Informed Consent Process Checklist to ensure that all participants receive the same information, have the opportunity to ask questions, and that study staff document that all required elements were explained. An Eligibility Confirmation Checklist will also be used to document each participant's eligibility prior to consent. The eligibility and consent process will occur either at the Day Report Center in a private location or at the Center for Rural and Community Health's (CRCH) Participant Welcome Center located at the West Virginia School of Osteopathic Medicine (WVSOM) Main Campus, Room B222. Participants will be given the opportunity to read the consent form themselves, with study staff available to answer questions. Case managers from the Day Report Program may accompany participants if available, but their presence is not required. All consents will be conducted privately and with the awareness of Day Report Program staff.

After enrollment, participants will complete monthly questionnaires for six months. The questionnaires capture recovery capital, social capital, and Day Report Program violations or interactions. A complete list of reportable Day Report Program violations can be found at: https://greenbriercounty.net/departments/day-report/. Questionnaires are administered in REDCap, a HIPAA-compliant survey platform commonly used in clinical trials. A description of the REC-CAP item list and scoring methodology was provided in the IRB submission and can be made available to regulatory authorities upon request; the full proprietary questionnaires themselves are not publicly available. Participants may be withdrawn from the study if they are removed from the Day Report Program, engage in violent or unsafe behavior with staff or partners, or under extenuating circumstances deemed appropriate by the PI or WVSOM IRB.

Study Procedures, Materials, and Potential Risk Regardless of assignment to the comparator arm (standard of care) or experimental arm (CRAFT program), the same data will be collected, consistent with the parallel-arm design. Data collection includes a baseline survey at enrollment followed by monthly surveys for five additional months (six months total follow-up).

Surveys will be administered by study staff to minimize differences in interpretation or reading ability. Each participant will be assigned a unique study identification number, which will appear on questionnaires, informed consent forms, and eligibility documents. Only the informed consent form will include both the participant's name and study ID.

Only the minimum necessary private health information will be collected. Survey data will be collected using REC-CAP instruments through the secure WVCTSI REDCap server. Tablets may be used for data entry. All electronic data will be linked only by study ID and stored on encrypted servers with access restricted to authorized study staff.

If a deviation occurs (e.g., missing eligibility document, incomplete consent, or missing questionnaire), study staff will document the issue using an After the Fact Change Form, consistent with IRB requirements. Weekly data validation spot checks will be conducted by the PI, Coordinator, Compliance Manager, or designated QI staff to ensure accuracy and integrity of study records.

This study poses no more than minimal to moderate risk to participants. Potential risks include discomfort when discussing substance use, recovery capital, social capital, or Day Report Program incidents/violations. There is also a transportation-related risk when traveling with Mountain Transit Authority drivers, addressed through insurance coverage and driver training. Confidentiality risks may arise if identifiable data were inadvertently disclosed, which could be harmful or embarrassing; these risks are mitigated through secure data handling and de-identification procedures. Self-reported relapse or overdose disclosed in study surveys will remain confidential with study staff and will not be reported to Day Report Program case managers, although participants remain subject to the routine monitoring protocols of the Day Report Program. Additional unforeseeable risks may also occur.

Informed Consent and Assent All recruitment procedures and materials will comply with the WVSOM IRB and HIPAA guidelines. Participants will be recruited exclusively from the Day Report Program, limited to adults (≥18 years) who are active clients. Day Report Program staff are not eligible.

Day Report Program case coordinators will first confirm participant interest before referring individuals to the research team. Flyers may be posted within the Day Report Center, and participants will also have the option to view a recruitment video describing the study purpose, risks, and benefits.

Interested participants will be contacted by study staff to review eligibility criteria and schedule a baseline visit. Informed consent will be obtained in a private location at either the Day Report Center or the WVSOM Center for Rural and Community Health (CRCH) Participant Welcome Center, Room B222. Participants will have the opportunity to read the consent form, and the Study Coordinator will use an Informed Consent Process Checklist to verify that all required elements are explained and understood. Case managers may accompany participants if available, but their presence is not required.

A signed copy of the consent form will be provided to each participant, with the original stored in a locked cabinet at the PI's office or the CRCH Welcome Center. Electronic copies will also be securely stored. Eligibility will be confirmed using documentation from the Day Report Program, with completion of a standardized eligibility checklist by study staff. Assent is not necessary since all participants are adults.

Protections Against Risk All study personnel will complete Human Subjects Research Training and Good Clinical Practice (GCP) CITI modules for Social and Behavioral Researchers prior to involvement in study activities. WVSOM IRB approval will be obtained to ensure compliance with federal and state regulations and institutional policies.

Study staff will ensure that participants understand study procedures before signing consent, emphasizing that participation is voluntary, refusal to enroll will not affect their involvement in the Day Report Program, and they may withdraw at any time without penalty.

Adverse events (AEs) may be reported directly by participants or by Day Report Program case managers. The Compliance Manager will complete AE, SAE, or Unanticipated Problem forms, which will then be reviewed and signed by the Principal Investigator (PI) prior to submission to the WVSOM IRB. Any serious or unexpected AE/UP will be reported to the IRB within 7 days of the study team becoming aware of the event. Monitoring of AEs will be performed by the PI and Compliance Manager, with weekly data validation spot reviews by the PI, Coordinator, or QI staff. If an AE suggests increased risk, the study team will re-evaluate study risk and document the issue using an After the Fact Change Form, along with required AE/SAE reports and IRB notification.

Data security procedures include storing completed hard-copy documents containing PHI in locked cabinets at the PI's office or CRCH Welcome Center (B222). Access to identifiable data is restricted to authorized study staff and regulatory authorities. Electronic data will be collected using REC-CAP through the secure WVCTSI REDCap server and stored on encrypted WVSOM CRCH servers. Identifiable violation data received from the Day Report Program will be replaced with study IDs and the originals securely destroyed. Identifiable data will otherwise be destroyed five years after study completion or three years after the last publication, whichever is later, unless regulations require longer retention.

Adverse events are defined as any undesirable sign, symptom, or medical condition occurring during the study or as a result of data collection. Serious adverse events (SAEs) include events that are fatal, life-threatening, require or prolong hospitalization, cause significant disability, or are otherwise judged serious by the investigator. Events will be graded as mild (no treatment required), moderate (resolved with treatment), or severe (inability to carry on normal activities and requiring professional care). Unanticipated problems are issues that increase risk to participants or others beyond what was previously known (e.g., a confidentiality breach causing serious social, legal, or economic harm).

Vulnerable Populations This study involves justice-involved adults. To protect this population, data collection will occur only in secure locations, either at the Day Report Center or within a private room on the WVSOM main campus. HIPAA safeguards are in place to maintain confidentiality and anonymity in the broader community context. Participants may be required to disclose to employers that they are enrolled in the Day Report Program or in other recovery-oriented services, or they may choose to self-disclose this information. Such information will not be shared beyond study staff and designated study partners (the Day Report Program, Jobs and Hope WV, and Mountain Transit Authority). These partners are noted in the informed consent as having access to participant data only as necessary to provide services.

Potential Benefits to Subjects and Others Benefits to participation include access to free transportation, cognitive behavioral therapy rewards overseen and provided by the Day Report Program, and employment support services. Multiple safeguards have been implemented to ensure participant safety. The findings of this study will provide important evidence for the public, medical providers, policymakers, and public health practitioners. The Substance Abuse and Mental Health Services Administration identifies gainful employment as a key predictor of long-term recovery and positive outcomes among individuals with a history of substance use.

Importance of Knowledge to Be Gained The knowledge to be gained from this study outweighs the potential risks, which are expected to be minimal. Multiple safeguards are in place to minimize risks as described above. This study will also lay the groundwork for future randomized clinical trials evaluating larger-scale, multi-center workforce models for recovery populations. Workforce development is critical to sustaining healthy communities. In states such as West Virginia, where a high proportion of the population are aging adults, stagnant workforce trends can lead to business closures and hinder economic development. This study explores innovative workforce models to support recovery while strengthening local economies.

ELIGIBILITY:
Inclusion Criteria:

* Active client of the Greenbrier County, West Virginia Day Report program.
* 18+ years of age
* An adult who has been charged with a nonviolent felony or misdemeanor offense and have a substance abuse problem.

Exclusion Criteria:

* Persons with a prior felony conviction in which he/she used force against another person with intent to cause serious bodily harm or death
* An offender is currently charged with a sexual offense or any offense involving a child victim or offense involving the illegal use of a firearm or other dangerous weapon.
* If death or serious bodily injury occurred to any person during an offender's crime or if any offender used force against another person during an offender's crime or if any offender used force against another person during the crime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in REC-CAP Social Capital Scale score from baseline to 6 months | 6 months
  Social recovery capital will be measured using the REC-CAP Social Recovery Capital Scale. Mean change in scores from baseline to 6 months will be compared between the CRAFT intervention group and the standard employment group.
Mean change in REC-CAP Recovery Capital Index score from baseline to 6 months | 6 months
  Personal recovery capital will be measured using the REC-CAP Recovery Capital Index. Mean change in scores from baseline to 6 months will be compared between the CRAFT intervention group and the standard employment group.
Number of reportable Day Report Program violations per participant over 6 months | 6 months
  Violations will be abstracted from Day Report Program records and summarized as the number of reportable incidents per participant. Mean monthly violations over 6 months will be compared between groups

SECONDARY OUTCOMES:
Sex-based differences in REC-CAP recovery capital scores and Day Report Program violations | 6 months
  Recovery capital scores (REC-CAP Social Recovery Capital and Recovery Capital Index) and number of Day Report Program violations will be analyzed by sex (male vs. female) to assess differential effects of the CRAFT workforce model.
Age-based differences in REC-CAP recovery capital scores and Day Report Program violations | 6 months
  Recovery capital scores (REC-CAP Social Recovery Capital and Recovery Capital Index) and number of Day Report Program violations will be analyzed by age group (18-29, 30-44, ≥45) to assess differential effects of the CRAFT workforce model.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Hendricks, PhD, Principal Investigator — WV School of Osteopathic Medicine
Locations (1):
- West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data and data dictionary
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon completion of the study and before primary publication. End date for sharing will be in accordance with institutional guidance and ICMJE recommendations.
Access Criteria: Upon request. Requests can be made through email to the study PI after the investigators have secured institutional board approval.